CLINICAL TRIAL: NCT05264311
Title: Effect of a Pilates Exercise Program on the Flexion-relaxation Rate in Women With Chronic
Brief Title: Pilates in Women With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marco Romagnoli, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-1292671
Record Dates: First submitted 2022-02-10; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Back Pain, Low
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EG: Exercise Group (Experimental): Pilates exercise program (1 h x 2 sessions per week x 2 months)
  Interventions: Other: Pilates exercise program
- CG: Control Group (No Intervention): Usual lifestyle

INTERVENTIONS:
Other: Pilates exercise program — The Pilates Exercise Program (PEP) (1 h x 2 sessions per week x 2 months) was delivered by one Pilates professional (with a mean of 6.5 years of experience in Pilates). The PEP carried out by Pilates instructor has been published in a previous study [31]. The exercises focused on core stability, posture, breathing, flexibility, strength, and muscle control, being the active awareness of the use of trunk muscles to stabilize the pelvic-lumbar region the main approach. The exercises performed were: the hundred, the rolled up, single leg circles with bent leg, spine stretch, rolling like a ball and single leg stretch. Each exercise was performed as follows: 4 repetitions of 30 seconds with 2 minutes of recovery between repetitions. In order to complete the 60 minutes session two exercises: the "superman" and the double leg bridge were added to the mentioned PEP.
  Other Names: Core strength exercise program
  Arms: EG: Exercise Group

SUMMARY:
The purpose of this study is to evaluate the effect of a Pilates exercise program (PEP) on the flexo-relaxation ratio (FRR) of the erector spinae (ES) muscle during standing maximal trunk flexion/extension in women with chronic low-back pain (LBP). A secondary goal is to investigate the effect of PEP on full trunk flexion ROM (TFRoM), pain intensity and functional capacity and analyse their relationship with the FRR.

DETAILED DESCRIPTION:
Purpose: To evaluate the effect of a Pilates exercise program (PEP) on the flexo-relaxation ratio (FRR) of the erector spinae (ES) muscle during standing maximal trunk flexion/extension in women with chronic low-back pain (LBP). A secondary goal was to investigate the effect of PEP on full trunk flexion ROM (TFRoM), pain intensity and functional capacity and analyse their relationship with the FRR. Material and methods: Thirty women with chronic LPB were randomly assigned to either PEP (EG, n=15) or control group (CG=15). EG followed an 8-week PEP while no specific intervention was carried out on the controls. Before and after this period all variables were recorded.

ELIGIBILITY:
Inclusion Criteria:

* lumbar or lumbosacral pain (with or without radicular pain) for at least six months;
* a score higher than 6/50 on the Oswestry Disability Index (ODI)
* absence of any back treatment for the last three months.

Exclusion Criteria:

* body mass index > 30 kg/m2
* prior surgery of the pelvis,
* spinal column or lower extremity
* scoliosis;
* systemic or degenerative disease
* history of neurological diseases or deficits not related to back pain
* pregnancy or hypertension.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
FRR was calculated by dividing the maximal EMG amplitude during flexion by the minimum EMG amplitude at full flexion. The mean of the 3 trials performed was used to determine the FRR for each muscle for each subject. | 2 months
  A lower FRR indicated a greater state of muscle relaxation. Asymmetry in muscle activity between both (right and left) ES muscles was calculated as their mean difference in RMS in the three flexion-extension tasks. Asymmetry in the FRR was calculated as the absolute difference between FRR of the right and left ES muscles.

SECONDARY OUTCOMES:
Full TFRoM was calculated as the average TFRoM from the three flexion-extension tasks. | 2 months
  To obtain the full trunk flexion ROM (TFRoM), the angular position of the inertial EMG sensor (attached with a kinesio-tape at T3 vertebrae) was measured from the start to the end of the flexion movement.
The version adapted to the Spanish population of the Low Back Outcome Score (LBOS) questionnaire was used to measure self-reported functional capacity. | 2 months
  LBOS was measured at pre-intervention (T0) and pos-intervention (T8).
A 10-cm Visual Analog Scale (VAS) was used to evaluate pain intensity | 2 months
  VAS was measured at pre-intervention (T0) and pos-intervention (T8).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ferri-Caruana, PhD, Principal Investigator — Department of Physical Activity and Sports. University of Valencia
Locations (1):
- Faculty of Physical Activity and Sport Sciences. University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No